CLINICAL TRIAL: NCT05224258
Title: Evaluation of the MiniMed™ 780G System in Type 1 Adult and Pediatric Subjects Utilizing Insulin Fiasp® (Insulin Aspart Injection)
Brief Title: Evaluation of the MiniMed™ 780G System in Type 1 Adult and Pediatric Subjects Utilizing Insulin Fiasp®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP336
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MiniMed 780G System Utilizing Insulin Fiasp (Experimental): Subjects with insulin-requiring type 1 diabetes age 7-80 using the MiniMed 780G system with Insulin Fiasp® for a period of three months.
  Interventions: Device: MiniMed 780G System

INTERVENTIONS:
Device: MiniMed 780G System — 780G System used with Insulin Fiasp® (Insulin Aspart Injection)

SUMMARY:
This global study (US, Canada, and Australia) will evaluate the safety and effectiveness of the MiniMed 780G system in type 1 adult and pediatric subjects utilizing Fiasp (insulin aspart injection) in a home setting.

DETAILED DESCRIPTION:
This global study is a multi-center, single arm study in insulin-requiring adult and pediatric subjects with type 1 diabetes on the MiniMed 780G system using Fiasp insulin as well as Medtronic Extended infusion set and reservoir. The run-in period and study period will be approximately 120 days long.

A total of up to 250 subjects with insulin-requiring type 1 diabetes age 7-80 will be enrolled at up to 25 investigational centers across the United States, Canada, and Australia in order to have 200 subjects enter the study period. Up to 125 subjects will be enrolled in the pediatric age group (7-17 years of age), up to 125 in the adult age group (18 years or older)

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age 7 - 80 years at time of screening.
2. Has a clinical diagnosis of type 1 diabetes:

   1. 14 - 80 years of age: A clinical diagnosis of type 1 diabetes for 2 years or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
   2. 7 - 13 years of age: A clinical diagnosis of type 1 diabetes for 1 year or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
3. Does not require a legally authorized representative to consent on their behalf due to mental or intellectual disability.
4. Subject or parent/caregiver is literate and able to read one of the languages offered in the pump.
5. Subject and/or legally authorized representative is willing to provide informed consent for participation.
6. Is willing to perform fingerstick blood glucose measurements as needed.
7. Is willing to wear the system continuously throughout the study.
8. Must have a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units and maximum total daily dose of 250 units or less.
9. Has a Glycosylated hemoglobin (HbA1c) less than 10% (as processed by Central Lab) at time of screening visit.

   Note: All HbA1c blood specimens will be sent to and tested by a National Glycohemoglobin Standardization Program (NGSP) certified Central Laboratory. HbA1c testing must follow NGSP standards.
10. Has thyroid-stimulating hormone (TSH) in the normal range OR if the TSH is out of normal reference range the Free T3 is below or within the lab's reference range and Free T4 is within the normal reference range.
11. Uses pump therapy for greater than 6 months prior to screening (with or without CGM experience)
12. Is willing to upload data from the study pump, must have Internet access, and a computer system, or compatible smartphone that meets the requirements for uploading the study pump.
13. Is willing to take one of the following insulins and can financially support the use of either of the 2 insulin preparations as required during the run-in period:

    1. Humalog (insulin lispro injection)
    2. NovoLog/NovoRapid (insulin aspart injection)
14. Is willing to take Fiasp insulin during the study period (supplied via Sponsor).

EXCLUSION CRITERIA:

1. Has hypersensitivity to insulin aspart or one of the excipients in Fiasp.
2. Has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to screening:

   1. Medical assistance (i.e., Paramedics, Emergency Room [ER] or Hospitalization)
   2. Coma
   3. Seizures
3. Has been hospitalized or has visited the ER in the 6 months prior to screening resulting in a primary diagnosis of uncontrolled diabetes.
4. Has had DKA in the last 6 months prior to screening visit.
5. Will not tolerate tape adhesive in the area of sensor placement as assessed by a qualified individual.
6. Has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
7. Is female of child-bearing potential and result of pregnancy test is positive at screening.
8. Is sexually active female of child-bearing potential and is not using a form of contraception deemed reliable by the investigator.
9. Is female and plans to become pregnant during the course of the study.
10. Is being treated for hyperthyroidism at time of screening.
11. Has diagnosis of adrenal insufficiency.
12. Has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.
13. Is using hydroxyurea at time of screening or plans to use it during the study.
14. Is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks.
15. Is currently abusing illicit drugs.
16. Is currently abusing marijuana.
17. Is currently abusing prescription drugs.
18. Is currently abusing alcohol.
19. Using pramlintide (Symlin), DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of screening.
20. Has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator.
21. Has elective surgery planned that requires general anesthesia during the course of the study.
22. Has sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening.
23. Plans to receive red blood cell transfusion or erythropoietin over the course of study participation.
24. Is diagnosed with current eating disorder such as anorexia or bulimia.
25. Has been diagnosed with chronic kidney disease that results in chronic anemia.
26. Has a hematocrit that is below the normal reference range of lab used.
27. Is on dialysis.
28. Has serum creatinine of >2 mg/dL.
29. Has celiac disease that is not adequately treated as determined by the investigator.
30. Has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, or ventricular rhythm disturbances.
31. Has had history of cardiovascular event 1 year or more from the time of screening without

    1. a normal EKG and stress test within 6 months prior to screening or during screening or
    2. clearance from a qualified physician prior to receiving the study devices if there is an abnormal EKG or stress test.
32. Has 3 or more cardiovascular risk factors listed below without a normal EKG within 6 months prior to screening or during screening or clearance from a qualified physician if there is an abnormal EKG:

    * Age >35 years
    * Type 1 diabetes of >15 years' duration
    * Presence of any additional risk factor for coronary artery disease
    * Presence of microvascular disease (proliferative retinopathy or nephropathy, including microalbuminuria)
    * Presence of peripheral vascular disease
    * Presence of autonomic neuropathy
33. Is a member of the research staff involved with the study.
34. Has used a MiniMed 780G pump prior to screening.

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Liljenquist, MD, Principal Investigator — Rocky Mountain Clinical Research; Mark Warren, MD, Principal Investigator — Physicians East; John Reed, MD, Principal Investigator — Endocrine Research Solutions; Frances Broyles, MD, Principal Investigator — Rainier Clinical Research Center; Dorothy Shulman, MD, Principal Investigator — University of South Florida; Bruce Bode, MD, Principal Investigator — Atlanta Diabetes Associates; Halis Akturk, MD, Principal Investigator — University of Colorado, Denver; Paul Norwood, MD, Principal Investigator — Valley Research; Carla Demeterco-Berggren, MD, Principal Investigator — Rady's Children's Hospital; Alexander Abitbol, MD, Principal Investigator — LMC Clinical Research; Daniele Pacaud, MD, Principal Investigator — Alberta Children's Hospital Research Institute; James Thrasher, MD, Principal Investigator — Medical Investigations, Inc.; Bhuvana Sunil, MD, Principal Investigator — MultiCare Institute for Research & Innovation; Mark Kipnes, MD, Principal Investigator — Diabetes and Glandular Disease Clinic, P.A.; Asheesh Dewan, MD, Principal Investigator — The Docs LLC; Barry Reiner, MD, Principal Investigator — Barry J Reiner MD LLC; Gnanagurudasan Prakasam, MD, Principal Investigator — Sutter Institute for Medical Research; Bruce King, MD, Principal Investigator — John Hunter Childrens Hospital
Locations (18):
- United States (15):
  - Medical Investigations, Inc., Little Rock, Arkansas
  - Valley Research, Fresno, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Rady's Children's Hospital, San Diego, California
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Barry J Reiner MD, LLC, Baltimore, Maryland
  - The Docs, LLC, Las Vegas, Nevada
  - Physicians East, Greenville, North Carolina
  - Diabetes and Glandular Disease Clinic, P.A., San Antonio, Texas
  - Rainier Clinical Research Center, Renton, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- John Hunter Childrens Hospital, New Lambton, New South Wales, Australia
- Canada (2):
  - Alberta Children's Hospital Research Institute, Calgary, Alberta
  - LMC Clinical Research, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 240 subjects (115 with age 7-17 and 125 with age 18-80) enrolled at the beginning, with 14 (5 with age 7-17 and 9 with age 18-80) screen failure, 3 subjects with age 7-17 early withdrawn prior the study period, 223 subjects (107 with age 7-17 and 116 with age 18-80) started the study and became the Intention to Treat Population.
Groups:
- Subjects 7-17 Years of Age: Subjects with insulin-requiring type 1 diabetes age 7-17 using the MiniMed 780G system with Insulin Fiasp® for a period of three months.
  MiniMed 780G System: 780G System used with Insulin Fiasp® (Insulin Aspart Injection)
- Subjects 18-80 Years of Age: Subjects with insulin-requiring type 1 diabetes age 18-80 using the MiniMed 780G system with Insulin Fiasp® for a period of three months.
  MiniMed 780G System: 780G System used with Insulin Fiasp® (Insulin Aspart Injection)
Period: Overall Study
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Started | 107 | 116
Completed | 103 | 112
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Parent/Guardian | 1 | 0
Not completed — Study Product No Longer in Use | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Deviation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention to Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age | Total
Number analyzed (Participants) | 107 | 116 | 223
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.0 (2.4) | 48.3 (14.5) | 31.9 (20.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 110
  Male | 51 | 62 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 3 | 19
  Not Hispanic or Latino | 82 | 113 | 195
  Unknown or Not Reported | 9 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 5 | 12
  White | 82 | 105 | 187
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 11 | 1 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.2 (4.5) | 29.3 (6.2) | 26.4 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint - Change in HbA1c
Description: The overall mean change in HbA1c from baseline to end of 3-month study period. Non-inferiority test.
Time Frame: 3 months
Population: Intention to Treat Population with available data. Three subjects aged 7-17 and two subjects aged 18-80 did not collect A1C at the end of the study period, so 104 subjects aged 7-17 and 114 subjects aged 18-80 were analyzed at end of study period and the change from baseline to end of study period.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 104 | 114
Percentage of HbA1c | -0.2 (0.7) | -0.4 (0.6)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Non-Inferiority — The overall mean change in HbA1c from baseline to end of 3-month study period. The mean change will be estimated and compared to a threshold of -0.38% with a margin of 0.4%; p < 0.001, t-test, 1 sided; Mean difference from baseline to exit = -0.2, 95% CI 2-sided [-0.4 to -0.1] — This is one arm study, the differences of HbA1c from baseline to exit were summarized for this endpoint
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Non-Inferiority — The overall mean change in HbA1c from baseline to end of 3-month study period. The mean change will be estimated and compared to a threshold of -0.5% with a margin of 0.4%; p < 0.001, Wilcoxon (Mann-Whitney); Mean difference from baseline to exit = -0.4, 95% CI 2-sided [-0.5 to -0.2] — This is one arm study, the differences of HbA1c from baseline to exit were summarized for this endpoint

2. Primary Outcome: Primary Effectiveness Endpoint - Percent of Time in Range (TIR 70-180 mg/dL [3.9 -10.0 mmol/L])
Description: The mean % of time in range (TIR 70-180 mg/dL [3.9 -10.0 mmol/L]). Non-inferiority test.
Time Frame: Last 6-7 weeks of 3-month study period
Population: Intention to Treat Population with available data. One subject aged 7-17 and three subjects aged 18-80 did not have enough SG points at the last 6-7 weeks of the study period, so 106 subjects aged 7-17 and 113 subjects aged 18-80 were analyzed at last 6-7 weeks of study period.
Measure: Mean (Standard Deviation); unit: Percentage of Time in Range (TIR 70-180)
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 106 | 113
Percentage of Time in Range (TIR 70-180) | 65.7 (11.3) | 77.1 (9.6)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Non-Inferiority — The mean % of time in range (TIR 70-180 mg/dL [3.9 -10.0 mmol/L]) will be estimated and compared to a threshold of 65.3% with a margin of 7.5% and a significance level of 0.025 (one-sided); p < 0.001, Wilcoxon (Mann-Whitney); Mean of Final Value = 65.7, 95% CI 2-sided [63.5 to 67.9] — This is one arm study, the Percent of Time in Range (TIR 70-180 mg/dL [3.9 -10.0 mmol/L]) from the last 6-7 weeks of 3 month study period was summarized for this endpoint
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Non-Inferiority — The mean % of time in range (TIR 70-180 mg/dL [3.9 -10.0 mmol/L]) will be estimated and compared to a threshold of 73.7% with a margin of 7.5% and a significance level of 0.025 (one-sided); p < 0.001, Wilcoxon (Mann-Whitney); Mean of Final Value = 77.1, 95% CI 2-sided [75.4 to 78.9] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Secondary Effectiveness Endpoint 1 - Percent of Time in Hypoglycemia (< 54 mg/dL [3.0 mmol/L])
Description: The mean % of time in hypoglycemia (< 54 mg/dL [3.0 mmol/L]). Non-inferiority test.
Time Frame: Last 6-7 weeks of 3 month study period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Time in Hypoglycemia (< 54
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 106 | 113
Percentage of Time in Hypoglycemia (< 54 | 0.3 (0.3) | 0.3 (0.4)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Non-Inferiority — The mean % of time in hypoglycemia (< 54 mg/dL [3.0 mmol/L]) will be estimated and compared to a threshold of 0.71% with a margin of 2% and a significance level of 0.025 (one-sided); p < 0.001, Wilcoxon (Mann-Whitney); Mean of Final Value = 0.3, 95% CI 2-sided [0.3 to 0.4] — This is one arm study, the Percent of Time in Hypoglycemia (< 54 mg/dL [3.0 mmol/L]) from the last 6-7 weeks of 3 month study period was summarized for this endpoint
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Non-Inferiority — The mean % of time in hypoglycemia (< 54 mg/dL [3.0 mmol/L]) will be estimated and compared to a threshold of 0.86% with a margin of 2% and a significance level of 0.025 (one-sided); p < 0.001, Wilcoxon (Mann-Whitney); Mean of Final Value = 0.3, 95% CI 2-sided [0.2 to 0.4] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Secondary Effectiveness Endpoint 2 - Percent of Time in Range (TIR 70-180 mg/dL [3.9 -10.0 mmol/L])
Description: The mean % of time in range (TIR 70-180 mg/dL [3.9 -10.0 mmol/L]).Superiority test.
Time Frame: Last 6-7 weeks of 3 month study period
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Time in Range (TIR 70-180)
Arm/Group | Subjects 7-17 Years of Age | Subjects 18-80 Years of Age
Number analyzed (Participants) | 106 | 113
Percentage of Time in Range (TIR 70-180) | 65.7 (11.3) | 77.1 (9.6)
Statistical Analysis 1: Comparison: Subjects 7-17 Years of Age; Test type: Superiority — The mean % of time in range (TIR 70-180 mg/dL [3.9 -10.0 mmol/L]) will be estimated and compared to a threshold of 65.3% and a significance level of 0.025 (one-sided); p = 0.208, Wilcoxon (Mann-Whitney); Mean of Final Value = 65.7, 95% CI 2-sided [63.5 to 67.9] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Subjects 18-80 Years of Age; Test type: Superiority — The mean % of time in range (TIR 70-180 mg/dL [3.9 -10.0 mmol/L]) will be estimated and compared to a threshold of 73.7% and a significance level of 0.025 (one-sided); p < 0.001, Wilcoxon (Mann-Whitney); Mean of Final Value = 77.1, 95% CI 2-sided [75.4 to 78.9] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 3-month Study Period
Description: Only Adverse Events during the study period were posted
Groups:
- Subjects 7-17 Years of Age Study Period: Subjects with insulin-requiring type 1 diabetes age 7-17 using the MiniMed 780G system with Insulin Fiasp® for a period of three months.
  MiniMed 780G System: 780G System used with Insulin Fiasp® (Insulin Aspart Injection)
- Subjects 18-80 Years of Age Study Period: Subjects with insulin-requiring type 1 diabetes age 18-80 using the MiniMed 780G system with Insulin Fiasp® for a period of three months.
  MiniMed 780G System: 780G System used with Insulin Fiasp® (Insulin Aspart Injection)
Arm/Group | Subjects 7-17 Years of Age Study Period | Subjects 18-80 Years of Age Study Period
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/116
Other Adverse Events (participants affected / at risk) | 26/107 | 30/116
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects 7-17 Years of Age Study Period (N=107) | Subjects 18-80 Years of Age Study Period (N=116)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Infusion site pain (General disorders) | 1 (3) | 0 (0)
Infusion site rash (General disorders) | 0 (0) | 1 (1)
Infusion site reaction (General disorders) | 1 (1) | 0 (0)
Medical device site irritation (General disorders) | 1 (1) | 0 (0)
Medical device site mass (General disorders) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 1 (1) | 1 (1)
Medical device site rash (General disorders) | 1 (2) | 2 (2)
Medical device site reaction (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Allergy to vaccine (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 5 (5)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Infusion site infection (Infections and infestations) | 3 (3) | 1 (1)
Medical device site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (3) | 1 (1)
Viral infection (Infections and infestations) | 4 (4) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acetonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT05224258/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05224258/SAP_001.pdf